CLINICAL TRIAL: NCT01266603
Title: A Phase II Trial of High Dose Interleukin-2 (HDIL-2) With Recombinant MAGE-A3 Protein Combined With Adjuvant System AS15 (recMAGE-A3 + AS15) in Patients With Unresectable or Metastatic Melanoma
Brief Title: High-Dose Interleukin-2 (HDIL-2), Combined With recMAGE-A3 + AS15 ASCI
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2010-0113; NCI-2011-00282 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2010-12-20; First posted 2010-12-24 (Estimated); Results first posted 2020-02-19 (Actual); Last update posted 2020-02-19 (Actual); Status verified 2020-02

CONDITIONS: Melanoma
Keywords: Metastatic Melanoma; Unresectable Melanoma; HDIL-2; Interleukin-2; IL-2; Aldesleukin; Proleukin; recMAGE-A3 + AS15; ASCI; recMAGE-A3; Recombinant MAGE-A3 protein; recMAGE-A3 + AS15 ASCI; MAGE-A3; MAGE-A3 ASCI
MeSH Terms: conditions — Melanoma | interventions — Interleukin-2; aldesleukin; MAGEA3 protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- HDIL-2 + recMAGE-A3 + AS15 (Experimental): HDIL-2 720,000 IU/kg by vein over an approximate 15 minute period every eight hours, for a maximum of 14 doses per cycle. recMAGE-A3 300 μg plus 420 μg of CpG7909 (a part of the Adjuvant System AS15) by intermuscular injection within 24 hours from first dose of HDIL-2.
  Interventions: Drug: HDIL-2; Biological: recMAGE-A3 + AS15

INTERVENTIONS:
Drug: HDIL-2 — 720,000 IU/kg by vein over an approximate 15 minute period every eight hours, for a maximum of 14 doses per cycle.
  Other Names: Interleukin-2; IL-2; Aldesleukin; Proleukin
Biological: recMAGE-A3 + AS15 — 300 μg plus 420 μg of CpG7909 (a part of the Adjuvant System AS15) by intermuscular injection within 24 hours from first dose of HDIL-2.
  Other Names: Recombinant MAGE-A3 Protein; recMAGE-A3 + AS15 ASCI; MAGE-A3; MAGE-A3 ASCI

SUMMARY:
The goal of this clinical research study is to learn if high-dose interleukin-2 (HDIL-2), when given in combination with recMAGE-A3 + AS15 ASCI (Antigen-Specific Cancer Immunotherapeutic), can help to control unresectable or metastatic melanoma in patients whose tumor tissue has the MAGE-A3 protein. The safety of this drug combination will also be studied. Researchers will also use samples of the original tumor or metastatic tissue (for example, lymph nodes or liver or lung) that are collected during screening to study if response to the study drug is related to the genes in the tissue.

DETAILED DESCRIPTION:
The Study Drugs:

HDIL-2 is similar to a hormone naturally found in the body that boosts the immune system by helping "natural killer" (NK) cells live longer and work better. NK cells are a type of white blood cell that kill other cells, and they may kill cancer cells.

ASCI is a immunotherapy designed to teach your immune system to fight cancer in the same way that you are given vaccines to prevent disease by teaching your immune system to fight an infection caused by germs. Because the cancer is made by your own body, the immune system does not recognize the cancer cells as being harmful. Your immune system needs to be "trained" to recognize the cancer cells. This is done by injecting a protein (the MAGE-A3 protein) that is found in the tumor and training your body to recognize it and to destroy the cells that have this protein. This may increase the effectiveness of IL-2 by slowing the growth of the cancer cells, which may cause them to die.

Study Drug Administration:

If you are found to be eligible to take part in this study, you will begin the study drugs within 14 days of signing the second consent form. To receive the study drugs, you will be admitted to the hospital, either in the intensive care unit (ICU) or a specifically designated nursing unit where study drugs can be administered, on Day 2 of each cycle and may remain in the hospital for up to 7 days each cycle.

You may receive a total of 24 ASCI doses either in combination with HDIL-2 or alone. You may receive the study drugs in combination for up to 30 weeks. After that, you may receive the ASCI study medication alone for up to 157 more weeks.

Cycle 1 is 14 days (Weeks 1 and 2):

* On Day 1 of Cycle 1, you will receive the ASCI study medication as an injection. Each injection will be given in the muscle of your upper arm or in your thigh. You will be watched in the clinic for at least 30 minutes after each injection.
* On Day 2 (+/- 2 business days), you will receive HDIL-2 through a catheter (a small plastic tube that is put into your vein under your collar bone or in your arm) over 15 minutes. HDIL-2 treatment will be delayed in cycles 2, 3, 4, 5, 6, 7, or 8 until all HDIL-2 related side effects either go away or the study doctor thinks they are under control.

Cycle 2 is 42 days (Weeks 3-8):

* On Day 1 of Weeks 3, 5, and 7 (+/- 2 business days) , you will receive the ASCI study medication as an injection.
* On Day 2 of Week 3 (+/- 2 business days), you will receive HDIL-2 by vein.

Cycle 3 is 14 days (Weeks 9 and 10):

* On Day 1 of Week 9 (+/- 2 business days), you will receive the ASCI study medication as an injection.
* On Day 2 of Week 9 (+/- 2 business days), you will receive HDIL-2 by vein.

Cycle 4 is 49 days (Weeks 11-17):

* On Day 1 of Weeks 11 and 15 (+/- 2 business days), you will receive the ASCI study medication as an injection.
* On Day 2 of Week 11 (+/- 2 business days), you will receive HDIL-2 by vein.

Cycle 5 is 21 days (Weeks 18-20):

* On Day 1 of Week 18 (+/- 2 business days), you will receive the ASCI study medication an injection.
* On Day 2 of Week 18 (+/- 2 business days), you will receive HDIL-2 by vein.

Cycle 6 is 42 days (Weeks 21-26):

* On Day 1 of Weeks 18, 21, and 24 (+/- 2 business days), you will receive the ASCI study medication as an injection.
* On Day 2 of Weeks 18 and 21 (+/- 2 business days), you will receive HDIL-2 by vein.

Cycle 7 is 21 days (Weeks 27-29):

* On Day 1 of Week 27 (+/- 2 business days), you will receive the ASCI study medication as an injection.
* On Day 2 of Week 27(+/- 2 business days), you will receive HDIL-2 by vein.

Cycle 8 is 28 days (Weeks 30-33):

* On Day 1 of Week 30 (+/- 2 business days), you will receive the ASCI study medication as an injection.
* On Day 2 of Week 30 (+/- 2 business days), you will receive HDIL-2 by vein.

On Day 1 of Weeks 34, 40, 46, 52, 64, 76, 88, and 100 (+/- 2 business days), you will receive the ASCI study medication as an injection.

Study Visits:

On Day 1 of Weeks 1, 3, 5, 7, 9, 11, 15, 18, 21, 24, 27, and 30 (+/- 2 business days):

* You will have a physical exam, including measurement of your weight and vital signs. °Blood (about 2 tablespoons) will be drawn for routine tests.
* You will be asked about any side effects you may be having and drugs you are taking.

On Day 2 of Weeks 1, 3, 5, 7, 9, 11, 18, 21, 27, and 30 (+/- 2 business days):

* Blood (about 2 tablespoons) will be drawn for routine tests.
* You will be asked about any side effects you may be having and drugs you are taking.

During Weeks 8, 17, 26, 33, 39, 51, 63, 75, 87, 99, 123, 147, 171, and 195 (+/- 1 week):

* You will have and a CT scan of your chest, abdomen, and pelvis to check the status of the disease.
* You will also have an MRI scan or CT scan of the brain to check the status of the disease.
* You will have photographs of your lesions taken if indicated by your doctor.

On Day 1 of Weeks 34, 40, 46, 52, 64, 76, 88, 100, 124, 148, 172, and 196 (+/- 2 business days):

* You will have a physical exam, including measurement of your weight and vital signs.
* Blood (about 2 tablespoons) will be drawn for routine tests.
* You will be asked about any side effects you may be having and drugs you are taking.

Additional Blood Draws:

Additional blood (about 4 tablespoons each time) will be drawn for laboratory tests to look at how the study drug combination may affect the immune system. These blood draws will be collected on Day 1 of cycle 1 and again during cycle 1 48 hours after the last dose of IL-2. Additional blood draws (about 4 tablespoons each time) will also Part of the blood drawn for these tests will be sent to GSK Biologicals (or a contracted laboratory) for testing.

Length of Study:

You may continue to receive the study drug combination for up to 8 cycles (33 weeks) and ASCI alone for up to 76 more weeks (+/- 2 business days). If you continue beyond completing 8 cycles of HDIL-2, you will receive the ASCI on Day 1 (+/- 2 business days) every 6 weeks for 4 doses (weeks 34, 50, 46, and 52), then on Day 1 (+/- 2 business days) every 12 weeks (weeks 64, 76, 98, and 110) for 4 doses, then on Day 1 (+/- 2 business days) of every 24 weeks (Weeks 134, 158, 182, and 187) for 4 doses.

You will be taken off the study therapy early if the disease gets worse, you experience intolerable side effects, or the study doctor thinks it is in your best interest. If you are removed from the study because of intolerable side effects, you will be followed weekly by either a phone call or clinic visit until the side effect is tolerable.

End-of-Dosing Visit:

After receiving the last dose of study drug combination, you will have an end-of-dosing visit:

* Your medical history will be reviewed and you will be asked about any side effects you may be having and drugs you are taking.
* You will have a physical exam, including measurement of your weight and vital signs.
* Blood (about 3 tablespoons) will be drawn for routine tests and ANA testing.

Follow-Up Visits:

You will have follow-up visits after your last dose of study drug, if the disease does not get any worse. Starting after the last dose of study drug, you will have 1 visit every 3 months for the 1st year, every 4 months for the 2nd year, every 6 months for the 3rd and 4th year, then once a year for up to 10 years (+/- 2 business days). At these visits, the following will be performed:

* You will have a physical exam, including measurement of your weight and vital signs.
* If the study doctor thinks it is needed, blood (about 2 tablespoons) will be drawn for routine tests.
* If the study doctor thinks it is needed, you will have a chest x-ray, CT scan of your chest, abdomen, and pelvis, and/or MRI scan or CT scan of the brain to check the status of the disease.

If the disease begins to get worse, information about the status of your health will be collected every 2 months. If you are not able to come into the clinic to complete this visit, you will be asked for this information over the phone. The phone call should last about 10-15 minutes each time.

This is an investigational study. IL-2 is commercially available and FDA approved for the treatment of metastatic melanoma. HDIL-2 is a higher dose than the standard approved dose of IL-2. The ASCI study medication is not FDA approved or commercially available. It is currently being used for research purposes only.

Up to 30 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. STEP 1 Written informed consent has been obtained from the patient before the performance of any protocol-specific procedure.
2. Male or female patient with histologically proven, measurable unresectable or metastatic cutaneous melanoma
3. Patient is >/= 18 years of age.
4. Formalin-fixed paraffin-embedded (FFPE) tumor tissue must be available for MAGE-A3 expression screening test from cutaneous, subcutaneous, lymph node lesion, lung or liver lesion. Archival FFPE tumor tissue can be provided for the MAGE-A3 screening test, as long as the FFPE tumor tissue was obtained from a biopsy or resection and no systemic chemotherapy, immunotherapy or targeted therapy has been received by the patient between the tumor collection and the MAGE-A3 screening test. Fresh tumor tissue in RNAlater must be also available for gene signature testing. Patients must have at least one biopsiable cutaneous, subcutaneous, lymph node lesion, The tumor sample should be preferably from the same lesion as the FFPE tumor tissue. Cutaneous lesions must measure >/= 4mm and lymph nodes, subcutaneous, lung or liver lesions must measure >/= 1cm.
5. STEP 2 ANA (antinuclear antibody) titer < 1:80
6. STEP 2 The patient's tumor shows expression of MAGE-A3 gene.
7. ECOG performance status of 0 or 1.
8. WBC >/= 3000/mm^3 and Hemoglobin >/= 9 g/dl
9. Platelet count >/= 100,000/mm^3.
10. Normal AST and ALT except for patients with liver metastases, in which serum ALT and AST </= 2.5 X upper limit of normal (ULN) will be permitted.
11. Creatinine </= 1.5 mg/dL
12. Normal total bilirubin except for patients with liver metastases, in which total bilirubin </= 1.5 X ULN will be permitted (patients with Gilbert's syndrome must have a total bilirubin less that 3.0 mg/dL).
13. LDH </= 2 X ULN
14. Stress cardiac test (stress thallium, stress MUGA, dobutamine echocardiogram or other stress test that will rule out cardiac ischemia) with estimated ejection fraction >50% within 6 months of signing consent form
15. Pulmonary function tests showing FEV1 > 65% or FVC > 65% of predicted within 6 months of signing consent form
16. Women of childbearing potential (WOCBP) must be using an adequate method of contraception prior to treatment, throughout the study, and for up to 8 weeks after the last dose of investigational product, in such a manner that the risk of pregnancy is minimized. In general, the decision for appropriate methods to prevent pregnancy should be determined by discussions between the investigator and the study subject. WOCBP include any female who has experienced menarche and who has not undergone successful surgical sterilization (hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or is not post-menopausal. Post-menopause is defined as: Amenorrhea for 12 consecutive months without another cause, or For women with irregular menstrual periods and taking hormone replacement therapy (HRT), a documented serum follicle stimulating hormone (FSH) level 35 mIU/mL.
17. (Continued #16) Women who are using oral contraceptives, other hormonal contraceptives (vaginal products, skin patches, or implanted or injectable products), or mechanical products such as an intrauterine device or barrier methods (diaphragm, condoms, spermicides) to prevent pregnancy, or are practicing abstinence or where their partner is sterile (eg, vasectomy) should be considered to be of childbearing potential. WOCBP must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 14 days before the start of treatment.
18. Men must also agree to use an adequate method of contraception.

Exclusion Criteria:

1. The patient has at any time received systemic chemotherapy, immunotherapy or targeted therapy (except for isolated limb perfusion, interferon, or radiation in the adjuvant setting, as long as this was performed at least 4 weeks before first study treatment administration).
2. Brain metastasis or history of brain metastasis.
3. Any types of melanoma other than cutaneous, i.e. ocular or mucosal .
4. The patient received any cancer immunotherapeutic containing a MAGE-A3 antigen.
5. Patients with a history of second malignancies are eligible provided that they have been free of recurrence from secondary malignancy for at least 3 years, does not include squamous cell carcinoma, basal cell carcinoma, or carcinoma in situ.
6. The patient has a history of an autoimmune disease such as, but not limited to, multiple sclerosis, lupus, rheumatoid arthritis, and inflammatory bowel disease or an antinuclear antibody (ANA) titer > 1:80.
7. The patient has a history of allergic disease or reactions likely to be exacerbated by any component of the study investigational compound.
8. The patient has a family history of congenital or hereditary immunodeficiency.
9. Known to be positive for viral hepatitis B or C (HBsAg or Anti HCV) or HIV (HIV antibodies) Patients should have a negative test within 6 months of starting treatment.
10. Systemic steroid therapy, steroid-containing compounds or any other immunosuppressive agents or to be used for more than 7 consecutive days (at a dose of prednisone or equivalent of >/= 0.125 mg/kg/day).
11. The patient has psychiatric or addictive disorders that may compromise his/her ability to give informed consent, or to comply with the trial procedures. Each patient will be evaluated by the principal investigator or his designee.
12. The patient has concurrent severe medical problems, unrelated to the malignancy, that would significantly limit full compliance with the study or expose the patient to unacceptable risk. Each patient will be evaluated by the principal investigator or his designee.
13. Initiation of another anti-cancer therapy.
14. For female patients: the patient is pregnant or lactating.
15. WOCBP who are unwilling or unable to use an acceptable contraceptive method to avoid pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2011-02-22 (Actual); Primary Completion 2018-11-01 (Actual); Study Completion 2018-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wen-Jen Hwu, MD,PHD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] McQuade JL, Homsi J, Torres-Cabala CA, Bassett R, Popuri RM, James ML, Vence LM, Hwu WJ. A phase II trial of recombinant MAGE-A3 protein with immunostimulant AS15 in combination with high-dose Interleukin-2 (HDIL2) induction therapy in metastatic melanoma. BMC Cancer. 2018 Dec 19;18(1):1274. doi: 10.1186/s12885-018-5193-9. PMID 30567529
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Groups:
- High-dose Interleukin-2 (HDIL-2) + recMAGE-A3 Protein (MAGE-A3: In the induction phase, 300 ug of MAGE-A3 +AS15 were given via intramuscular injection every 2 weeks for 6 cycles and then every 3 weeks for 6 cycles. HDIL-2 was initiated on the day following MAGE-A3 CI immunization or up to eight cycles on weeks 1,3,9,11,18.21,27 and 30 at 720,000 IU/kg every 8 h for up to 14 doses each cycle. Following completion of of the 30-week induction HDIL-2 + MAGE-A3, patients who remained on study were continued on the maintenance MAGE-A3 alone alone given every 6 weeks for 4 cycles, then every 12 weeks for 4 cycles, and then every 24 weeks for 4 cycles.
Period: Overall Study
Arm/Group | High-dose Interleukin-2 (HDIL-2) + recMAGE-A3 Protein (MAGE-A3
Started | 44
MAGE-A3 Positive Tumor | 18
Patients Evaluable for Safety | 17
Patients Evaluable for Response | 16
Continued to Maintenance- MAGE-A3 | 4
Maintenance Completion | 2
Completed | 2
Not Completed | 42
Not completed — Adverse Event | 1
Not completed — Lack of Efficacy | 14
Not completed — Withdrawal by Subject | 1
Not completed — Failed screening; MAGE-A3 negative | 26

BASELINE CHARACTERISTICS:
Arm/Group | High-dose Interleukin-2 (HDIL-2) + recMAGE-A3 Protein (MAGE-A3
Number analyzed (Participants) | 17
Age, Continuous [Mean (Full Range); unit: Years] | 55 [30 to 64]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 17
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 17
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 17

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate
Description: To evaluate the objective response rate induced by the concurrent administration of HDIL-2 and recMAGE-A3 + AS15 ASCI in patients with MAGE-A3-positive, unresectable or metastatic melanoma. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: Until disease progression or up to 3 years & 9 months
Measure: Number; unit: percentage of participants
Arm/Group | High-dose Interleukin-2 (HDIL-2) + recMAGE-A3 Protein (MAGE-A3
Number analyzed (Participants) | 16
percentage of participants | 25

2. Secondary Outcome: Rate of SAEs
Description: To evaluate the safety and toxicity profile of HDIL-2 in combination with recMAGE-A3 + AS15 ASCI in participants with MAGE-A3-positive, unresectable or metastatic melanoma
Time Frame: Until treatment completed or up to 3 years & 9 months
Measure: Number; unit: participants
Arm/Group | High-dose Interleukin-2 (HDIL-2) + recMAGE-A3 Protein (MAGE-A3
Number analyzed (Participants) | 17
participants | 1

3. Secondary Outcome: Progression-free Survival
Description: To evaluate the rate of stable disease, progression-free survival and the overall survival of patients with MAGE-A3- positive, unresectable or metastatic melanoma who received the combination of HDIL-2 and recMAGE-A3 + AS15 ASCI.
Time Frame: Until treatment completed or up to 3 years & 9 months.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | High-dose Interleukin-2 (HDIL-2) + recMAGE-A3 Protein (MAGE-A3
Number analyzed (Participants) | 17
Months | 3.6 [1.8 to 12]

ADVERSE EVENTS:
Time Frame: Throughout treatment up to 3 years & 9 months.
Arm/Group | High-dose Interleukin-2 (HDIL-2) + recMAGE-A3 Protein (MAGE-A3
All-Cause Mortality (participants affected / at risk) | 5/17
Serious Adverse Events (participants affected / at risk) | 1/17
Other Adverse Events (participants affected / at risk) | 17/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | High-dose Interleukin-2 (HDIL-2) + recMAGE-A3 Protein (MAGE-A3 (N=17)
Renal Insufficiency (Renal and urinary disorders) | 1
Hyperuricemia (Metabolism and nutrition disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Hypothyroidism (Endocrine disorders) | 1
Hypotension (Cardiac disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 1
Ventricular Tachycardia (Cardiac disorders) | 1
Gastroperesis (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | High-dose Interleukin-2 (HDIL-2) + recMAGE-A3 Protein (MAGE-A3 (N=17)
Anemia (Blood and lymphatic system disorders) | 14
Anorexia (Metabolism and nutrition disorders) | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 7
Chills (General disorders) | 10
Constipation (Gastrointestinal disorders) | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Decreased Urinary Output (Renal and urinary disorders) | 1
Diarrhea (Gastrointestinal disorders) | 7
Dry Skin (Skin and subcutaneous tissue disorders) | 15
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3
Edema (General disorders) | 14
Fatigue (General disorders) | 14
Fever (General disorders) | 5
Headache (Nervous system disorders) | 7
Hyperglycemia (Metabolism and nutrition disorders) | 6
Hyperkalemia (Metabolism and nutrition disorders) | 4
Hypermagenesemia (Metabolism and nutrition disorders) | 1
Hypertension (Vascular disorders) | 2
Hyperuricemia (Metabolism and nutrition disorders) | 4
Hypoalbunemia (Metabolism and nutrition disorders) | 14
Hypoglycemia (Metabolism and nutrition disorders) | 5
Hyponatremia (Metabolism and nutrition disorders) | 2
Hypophosphatemia (Metabolism and nutrition disorders) | 3
Hypotension (Vascular disorders) | 7
Increased Alanine Aminotransferase (Investigations) | 3
Increased Alkaline Phosphatase (Investigations) | 3
Increased Aspartate Aminotransferase (Investigations) | 5
Increased Bilirrubin (Investigations) | 6
Increased Creatinine (Renal and urinary disorders) | 6
Injection Site Reaction (General disorders) | 5
Lymphopenia (Investigations) | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 10
Nausea (Gastrointestinal disorders) | 11
Pain (Skin and subcutaneous tissue disorders) | 12
Peripheral Sensory Neuropathy (Nervous system disorders) | 7
Pruritis (Skin and subcutaneous tissue disorders) | 12
Rash (Skin and subcutaneous tissue disorders) | 8
Thrombocytopenia (Investigations) | 2
Tinnitus (Ear and labyrinth disorders) | 3
Ventricular tachycardia (Cardiac disorders) | 2
Vomiting (Gastrointestinal disorders) | 7
Weight Loss (Investigations) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-12-09): https://cdn.clinicaltrials.gov/large-docs/03/NCT01266603/Prot_SAP_000.pdf